CLINICAL TRIAL: NCT04850846
Title: A Randomized Placebo-Controlled Phase 2 Study of Metformin for the Prevention of Progression of Monoclonal Gammopathy of Undetermined Significance and Smoldering Multiple Myeloma
Brief Title: Investigation of Metformin for the Prevention of Progression of Precursor Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Omar Nadeem, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21-008; K22CA251648 (NIH)
Record Dates: First submitted 2021-03-18; First posted 2021-04-20 (Actual); Results first posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Monoclonal Gammopathy of Undetermined Significance; Smoldering Multiple Myeloma
Keywords: Monoclonal Gammopathy of Undetermined Significance; Smoldering Multiple Myeloma
MeSH Terms: conditions — Monoclonal Gammopathy of Undetermined Significance; Smoldering Multiple Myeloma | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Metformin (Experimental): Randomly assigned participants receive a stepped dose escalation until target daily dose of 1500mg Metformin XR is reached (3 x 500mg pills/day). The intervention duration will last an additional 6 months.
  Metformin Extension:
  Participants will have the option of unblinding at the end of their 6months treatment and those who were randomly assigned to the metformin experimental arm can continue taking metformin if they opt in. The extended intervention duration will last an additional 6 months. (1500mg Metformin XR or highest tolerated dose )
  Interventions: Drug: Metformin XR
- Placebo (Experimental): Randomly assigned participants receive a stepped dose escalation until target daily dose of 3 pills/day is reached. The intervention duration will last 6 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Metformin XR — Orally by mouth
  Other Names: Glucophage XR
  Arms: Metformin
Other: Placebo — Orally by mouth
  Arms: Placebo

SUMMARY:
The purpose of this research is to understand whether the drug metformin could be used in the future to help prevent patients with monoclonal gammopathy of undetermined significance (MGUS) and smoldering multiple myeloma (SMM) from developing multiple myeloma.

The names of the study drug involved in this study is:

* Metformin, extended release
* Placebo ( a pill that has no active ingredients)

DETAILED DESCRIPTION:
This is a Phase 2, double-blind, randomized placebo-controlled trial in patients with higher-risk monoclonal gammopathy of undetermined significance (MGUS) and low-risk smoldering multiple myeloma (SMM) to test the efficacy of metformin in reducing clinical indicators of disease progression in MGUS and SMM patients.

Metformin is considered "investigational", which means it has not been approved for the study of cancer prevention by the United States Food and Drug Administration. It has been approved for other uses including for blood sugar control in some people with Type II diabetes.

Multiple myeloma is a cancer of the plasma cells, which is an important part of the immune system. Patients with active multiple myeloma generally require treatment. There are currently no approved therapies for MGUS and SMM patients.

Metformin is a medication that is commonly used in the treatment of diabetes. Metformin works by decreasing glucose production in the liver, decreasing glucose absorption, and improving insulin sensitivity. This study is interested in studying this medication because several recent studies indicate that the drug may help prevent progression in patients with MGUS or SMM. This study is looking to learn more about whether metformin will benefit patients with MGUS or SMM who may not have diabetes.

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

After enrollment participants will be randomized assigned to receive either the Placebo or Metformin pills and to take them for 6 months depending on participant tolerance to the drug.

Participants will have the option to learn their treatment assignment after primary (6-month) outcome assessments are complete, and individuals randomized to metformin will have the opportunity to continue to take metformin for an additional 6-months to allow for the observation of potentially longer-term treatment response. Participants who choose to be unblinded and are taking placebo will discontinue study medication.

It is expected that about 80 people will take part in this research study.

The National Cancer Institute of the National Institutes of Health is supporting this trial.

ELIGIBILITY:
Inclusion Criteria:

-Diagnosed with higher-risk MGUS or low-risk SMM defined below:

--Higher-Risk MGUS: bone marrow plasma cell concentration <10%# AND either serum M-protein level ≥1.5 g/dL to <3 g/dL or abnormal free light-chain (FLC) ratio (<0.26 or>1.65) or IgA MGUS.

Note: individuals with an abnormal FLC ratio that are classified as light-chain only are eligible. Light-chain only patients are defined as complete loss of immunoglobulin heavy-chain, accompanied by abnormal FLC ratio with an increased level of the appropriate involved light-chain (increased kappa FLC in patient with ratio >1.65, and increased lambda FLC in patients with ratio <0.26).

* Low-Risk Smoldering Myeloma: bone marrow plasma cells ≥10%# with the absence of additional high-risk features, which are further defined in the exclusion criteria

  #A new bone marrow biopsy is preferred for plasma cell determination at screening; however, determination of eligibility can be made from most recent bone marrow biopsy performed as long as it was within 2 years of enrollment.
  * Absence of evidence of CRAB criteria* or new criteria of active MM or active WM which including the following (note if one or more criteria has not been evaluated (e.g., no MRI), the criteria for active MM or WM for that feature is considered unmet):
* Increased calcium levels (corrected serum calcium >0.25 mmol/dL above the upper limit of normal or >.275 mmol/dL) related to MM
* Renal insufficiency (attributable to MM)
* Anemia (Hb 2g/dL below the lower limit of normal or <10g/dL) related to MM
* Bone lesions (lytic lesions or generalized osteoporosis with compression fractures)
* Bone marrow plasma cells ≥60%
* Serum involved/uninvolved FLC ratio ≥100, provided the absolute level of the involved free light chain is at least 100 mg/L and repeated twice (light chain smoldering myeloma as described in section 2.4 is not an exclusion criteria).
* MRI with two or more focal lesion that is at least 5 mm or greater in size

  *Participants with CRAB criteria that are attributable to conditions other than the disease under study may be eligible
  * At least 18 years of age.
  * Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
  * The following laboratory values obtained prior to the first dose of study drug/placebo:
* AST and ALT < 1.5 x institutional ULN
* Serum bilirubin < institutional ULN (in patients with Gilbert's Disease, direct bilirubin < institutional ULN)
* Calculated creatinine clearance ≥ 45 mL/min

  * Estimation of renal function will be assessed using the CrCl calculated based on the Cockcroft-Gault formula:
  * CrCl (mL/min) = (140-age) (weight [kg]/72 (serum creatinine [mg/dL]; for females the formula is multiplied by 0.85
* Random glucose < 160 mg/dL or fasting glucose < 126 mg/dL (other values require workup to rule out undiagnosed diabetes that may require treatment)

  * Ability to understand and the willingness to sign a written informed consent document
  * For participants who wish to enroll in the open label extended treatment (crossover arm), participants can be unblinded and learn of their drug group AFTER completing primary endpoint collection. Patient must be randomized to metformin in order to continue taking metformin for 6 additional months.

Exclusion Criteria:

* Presence of high-risk smoldering myeloma, as defined by per IMWG/Mayo 2018 "20-2-20" Criteria (at least 2 of the following)

  * Bone marrow plasmacytosis ≥20%
  * ≥2g/dl M protein
  * ≥20 involved: uninvolved serum free light chain ratio
* Diagnosed or treated for another malignancy within the study period.
* Currently on medications for diabetes treatment

  * Patients with hyperglycemia (random glucose < 160 mg/dL or fasting glucose < 126 mg/dl) but who are not on any drug treatment are eligible
* Participants who are receiving any other investigational agents.
* Women who are pregnant or who are unable or unwilling to use contraception during the study period are excluded from this study because it is a class B agent which is known to cross the placenta rapidly and is unbound in serum.
* Any condition associated with increased risk of metformin-associated lactic acidosis (prior renal failure or liver failure, history of acidosis of any type) or habitual intake of 3 or more alcoholic beverages per day.
* Known intolerance to metformin
* Known malabsorption syndrome or diagnosis with a medical condition that may alter gastrointestinal absorption of medications including but not limited to inflammatory bowel disease impacting the small intestine or recent history of bariatric surgery.
* Any other condition that, in the investigator's judgment, would contraindicate the use of metformin or otherwise interfere with participation in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2025-01-29 (Actual); Study Completion 2027-07-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Omar Nadeem, MD, Principal Investigator — Dana-Farber Cancer Institute; Catherine R Marinac, PhD, Study Director — Dana-Farber Cancer Institute
Locations (7):
- United States (7):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber at Brighton, Brighton, Massachusetts
  - Dana-Farber at Merrimack Valley, Methuen, Massachusetts
  - Dana-Farber at Milford, Milford, Massachusetts
  - DF/ BWCC in Clinical Affiliation with South Shore Hospital, Weymouth, Massachusetts
  - Dana-Farber at NHOH, Londonderry, New Hampshire

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: CatherineR_Marinac@dfci.harvard.edu. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Metformin: Randomly assigned participants receive a stepped dose escalation until target daily dose of 1500mg Metformin XR is reached (3 x 500mg pills/day). The intervention duration will last an additional 6 months.
  Metformin Extension:
  Participants will have the option of unblinding at the end of their 6months treatment and those who were randomly assigned to the metformin experimental arm can continue taking metformin if they opt in. The extended intervention duration will last an additional 6 months. (1500mg Metformin XR or highest tolerated dose )
  Metformin XR: Orally by mouth
Period: Overall Study
Arm/Group | Metformin | Placebo
Started | 30 | 30
Completed | 22 | 23
Not Completed | 8 | 7
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Adverse Event | 3 | 1
Not completed — Subject stopped taking medication | 2 | 4
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Median (Full Range); unit: years] | 65 [38 to 80] | 65 [34 to 89] | 65 [34 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 14 | 16 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 29 | 29 | 58
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 26 | 25 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60
Diagnosis [Count of Participants; unit: Participants]
  MGUS | 11 | 12 | 23
  SMM | 19 | 18 | 37

OUTCOME MEASURES:

1. Primary Outcome: (M-)Protein Concentrations Change
Description: Assessed by using the serum-protein electrophoresis
Time Frame: Baseline to 6-months
Population: 8 participants in the metformin arm and 6 participants in the control arm did not have analyzable m-protein data.
Measure: Median (Full Range); unit: percent change
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 22 | 24
percent change | -3.2 [-33.0 to 20.4] | 7.7 [-15.4 to 29.7]

2. Secondary Outcome: Serum Free Light Chains Change by Mass Spectrometry
Time Frame: Baseline to 6-months
Reporting Status: Not Posted

3. Secondary Outcome: Hemoglobin Concentrations Change
Time Frame: Baseline to 6-months
Reporting Status: Not Posted

4. Secondary Outcome: Hemoglobin A1c (HbA1c) Concentrations Change
Time Frame: Baseline to 6-months
Reporting Status: Not Posted

5. Secondary Outcome: Molecular Evolution of CD138+ Cells
Time Frame: Baseline to 6-months
Reporting Status: Not Posted

6. Secondary Outcome: Molecular Evolution of Immune Cells (CD138- or CD45+)
Time Frame: Baseline to 6-months
Reporting Status: Not Posted

7. Secondary Outcome: Changes in Plasma Metabolites Measured by Liquid Chromatography-mass Spectrometry
Time Frame: Baseline to 6-months
Reporting Status: Not Posted

8. Secondary Outcome: Changes in PROMIS Global Health Summary Score v1.2
Time Frame: Baseline to 6-months
Reporting Status: Not Posted

9. Secondary Outcome: Number of Participants Willing to Continue to Take Metformin Beyond 6 Month Primary Assessment Period
Time Frame: Baseline- 12 months
Reporting Status: Not Posted

10. Secondary Outcome: Changes in Response for Those Who Choose to Take Metformin for up to 1 Year Per IMWG Response Criteria
Time Frame: Baseline- 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent, through 30 days after the last dose of study drug, up to 7 months for the initial randomized placebo-controlled phase and up to 13 months for participants who continued onto the extension phase
Arm/Group | Metformin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 1/30
Serious Adverse Events (participants affected / at risk) | 1/30 | 1/30
Other Adverse Events (participants affected / at risk) | 26/30 | 18/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=30) | Placebo (N=30)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1) | 0
Sepsis (Infections and infestations) | 0 | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin (N=30) | Placebo (N=30)
Nausea (Gastrointestinal disorders) | 14 | 9
Diarrhea (Gastrointestinal disorders) | 14 | 5
Constipation (Gastrointestinal disorders) | 8 | 3
Headache (Nervous system disorders) | 6 | 5
Bloating (Gastrointestinal disorders) | 8 | 2
Flatulence (Gastrointestinal disorders) | 4 | 4
Anorexia (Metabolism and nutrition disorders) | 6 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 2 | 3
Fatigue (General disorders) | 3 | 1
Creatinine increased (Investigations) | 2 | 1
Dizziness (Nervous system disorders) | 2 | 1
Dysgeusia (Nervous system disorders) | 2 | 1
Weight loss (Investigations) | 3 | 0
Belching (Gastrointestinal disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-06): https://cdn.clinicaltrials.gov/large-docs/46/NCT04850846/Prot_SAP_000.pdf